CLINICAL TRIAL: NCT01008748
Title: Determinants of Smoking Cessation Among Latinos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Department of Health and Human Services (U.S. Federal Agency); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0442; 2P60MD000503-05 (NIH)
Record Dates: First submitted 2009-10-02; First posted 2009-11-06 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Smoking Cessation
Keywords: Smoking; Latinos; Mexican American; Spanish-speaking smokers; Ecological momentary assessment; Nicotine patch; Smoking cessation counseling; Questionnaire; EMA
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Nicotine Replacement Therapy; Surveys and Questionnaires; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smoking Cessation Treatment (Experimental): Nicotine replacement therapy (NRT), self-help materials, + brief in-person and telephone counseling, all conducted in Spanish. Computerized questionnaires at each of 5 visits and will take 1 1/2 hours to complete each time.
  Interventions: Drug: Nicotine Replacement Therapy (NRT); Behavioral: Questionnaire; Behavioral: Counseling; Behavioral: Self-Help Materials

INTERVENTIONS:
Drug: Nicotine Replacement Therapy (NRT) — NRT for participants who smoke >10 cigarettes/day will consist of 2 weeks of 21 mg nicotine patches, 1 week of 14 mg patches, and 1 week of 7 mg patches. Nicotine Patch therapy for participants who smoke 5-10 cigarettes/day will consist of 2 weeks of 14 mg patches and 2 weeks of 7 mg patches. Patch dispensation will occur at weekly treatment visits.
  Other Names: Nicotine Patch Therapy
Behavioral: Questionnaire — Computerized questionnaires at each of 5 visits and will take 1 1/2 hours to complete each time.
  Other Names: Survey
Behavioral: Counseling — Each counseling session, whether face-to-face or over the phone, will last approximately 15 minutes. In-person counseling sessions occur at weeks -1, 0, and 3, with telephone counseling sessions occurring at weeks 0.5, 1, and 2. Counselors will conduct all sessions in Spanish.
Behavioral: Self-Help Materials — Spanish-language self-help materials currently used by the NCI's Cancer Information Service.
  Other Names: pamphlets

SUMMARY:
The goal of this study is to learn how neighborhood and individual factors affect the ability to stop smoking among Spanish-speaking Mexican American (MA) smokers who want to quit smoking.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will receive treatment to help you quit smoking, including written self-help materials, counseling, and a supply of the nicotine patch for 4 weeks. Over the next 6 months, you will visit M. D. Anderson 5 times during this study. You will also be called 3 times for smoking cessation counseling during this study.

Study Visits:

First (Orientation) Visit You will be asked about your feelings and moods, as well as how many cigarettes you smoke. You will fill out questionnaires on a computer. The questionnaires will be about your mood, stress level, and smoking-related issues. They should take about 1 hour and 30 minutes to complete.

You will complete a breath test. For the breath test, you will blow into a tube that's attached to a machine that is used to estimate the amount of tobacco smoke that you inhale.

You will give two saliva samples at this visit. To collect the first saliva sample, you will place a piece of cotton in your mouth for 3 minutes. The saliva sample is used to check the amount of cotinine in the body. Cotinine is a chemical that is produced in your saliva when your body breaks down nicotine.

The second saliva sample will be collected by spitting into a container. Researchers will perform genetic tests with these samples to look for genes that control the production and use of neurotransmitters, naturally occurring chemical messengers in the brain. People with certain genes may have a more difficult time quitting smoking, because of the way nicotine affects these chemicals. Your second saliva sample will be stored in a biorepository at M. D. Anderson for use in future research related to nicotine addiction, smoking, and/or cancer. Your saliva sample will be placed in a bank of biological samples and data that is available to researchers conducting research related to cancer or nicotine dependence.

Before your saliva sample can be used for research, the people doing the research must get specific approval from the Institutional Review Board (IRB) of M. D. Anderson. The IRB is a committee made up of doctors, researchers, and members of the community. The IRB is responsible for protecting the participants involved in research studies and making sure all research is done in a safe and ethical manner. All research done at M. D. Anderson, including research involving your saliva sample from this bank, must first be approved by the IRB.

Your samples will be given a code number. No identifying information will be directly linked to your samples. Only the researcher in charge of the bank will have access to the code numbers and be able to link the samples to you. Other researchers using your samples will not be able to link this data to you.

Genetic information obtained will not be provided to you.

Second (Baseline) Visit:

Your second visit (Baseline) will occur 1 week before your Quit date visit. You will fill out questionnaires on a computer. The questionnaires will be about your, stress level, social support and smoking-related issues. They should take about 1 hour and 30 minutes to complete.

You will complete a breath test. For the breath test, you will blow into a tube that's attached to a machine that is used to estimate the amount of tobacco smoke that you inhale.

Your Height, Weight and Waist circumference measures will be taken.

You will also receive individual counseling. During counseling, you will discuss techniques to help you quit smoking.

In addition, you will receive a small, hand-held personal computer and be trained in how to use it. You will carry this computer with you for 4 weeks. You will use the computer to answer questions about your mood, stress, and smoking-related issues. You will be asked to fill out some questions on the computer each time you have an urge to smoke or you actually smoke. Also, the computer will "beep" at random and set times and request that you answer some questions. This computer will not wake you during the night and you will be able to wait to answer questions for a few minutes if it goes off when you are busy. Answering the questions should take about 5 to 10 minutes.

Third (Quit Day) and Fourth (Week 3) Study Visits:

Your Third visit (Quit Day) will occur 1 week after your Second (Baseline) visit. Your Fourth visit will occur 3 weeks after your Quit Day. During these visits, you will be asked to fill out questionnaires on a computer about your moods and feelings, as well as how many cigarettes you smoke. The questionnaires should take about 30 minutes to complete.

You will also receive individual counseling. During counseling, you will discuss techniques to help you quit smoking.

On your Third visit, you will complete the breath test and your Weight and Waist circumference measures will also be taken.

At your Third visit you will be given a supply of nicotine patches to last until your Fourth visit.

At your Fourth visit you will be given a one week supply of nicotine patches. You will be on nicotine patches for a total of 4 weeks. At the Fourth Visit, you will also complete the breath test, will give a saliva sample and your Weight and Waist circumference measures will be taken.

Last (Week 26) Visit:

This visit will occur 26 weeks (or 6 months) after your Quit Day. During these visits, you will be asked to fill out questionnaires on a computer about your moods and feelings, as well as how many cigarettes you smoke.

The questionnaires should take about 1 1/2 hours to complete.

You will complete the breath test, your Weight and Waist circumference measures will be taken and you will also give a saliva sample at the last (Week 26) visit.

Telephone Calls:

Between your first (Orientation) visit and your Fourth (Week 3) visit, you will receive 3 calls from a smoking cessation counselor. You will receive your first call a few days before your quit day. You will receive a second call 1 week after your Quit Day and another call 2 weeks after your Quit Day. During these calls, you will discuss techniques to help you quit smoking. These calls will last 10 to 15 minutes and will be scheduled in advance.

Additional Information:

You may be contacted by mail, telephone, and/or e-mail throughout the study to remind you about clinic visits. You may also be asked for information about your smoking status during the usual reminder calls and/or calls to reschedule missed appointments.

Length of Study:

You will be considered off study when you complete the Week 26 (or Last) visit.

This is an investigational study. The nicotine patch is FDA approved and commercially available. Up to 200 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Current daily smoker who average >/= 5 cigarettes/day for the last year
2. Mexican-American (MA) Adults from the Houston-based MA Cohort Study and/or from the community
3. Age 18 to 65 years
4. Motivated to quit smoking in the next 30 days
5. Viable (working) telephone number and home address
6. Prefers to speak in Spanish
7. Register "8" or more on a carbon monoxide breath test

Exclusion Criteria:

1. Contraindication for nicotine patch use
2. Regular use of tobacco products other than cigarettes (cigars, pipes, smokeless tobacco)
3. Use of nicotine replacement therapy products or other smoking cessation medications, other than the nicotine patches supplied during the study
4. Pregnancy or lactation
5. Currently enrolled in a smoking cessation program
6. Participation in a smoking cessation program or study during the past 90 days
7. Another household member is enrolled in this protocol
8. Active substance abuse problem

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wetter, PhD, MS, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Vinci C, Cambron C, Lam C, Wetter DW. Perceived discrimination and smoking lapse among Mexican Americans: An ecological momentary assessment study. Health Psychol. 2021 Jun;40(6):388-397. doi: 10.1037/hea0001093. PMID 34323541
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 2009 and September 2016. Participants were recruited from the Mexican-American Cohort study and from Houston area.
Groups:
- Smoking Cessation Treatment: 6 wks of nicotine patch therapy, self-help guide and in-person/telephone individual counseling (6 sessions in 26 weeks) based on Tobacco Use and Dependence Clinical Practice Guideline
Period: Overall Study
Arm/Group | Smoking Cessation Treatment
Started | 200
Baseline | 188
Week 0 | 182
Week 3 | 168
Week 26 | 119
Completed | 119
Not Completed | 81
Not completed — Lost to Follow-up | 80
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Groups:
- Smoking Cessation Treatment: NRT, self-help materials + brief in-person and telephone counseling, all conducted in Spanish. Computerized questionnaires at each of 5 visits.
Arm/Group | Smoking Cessation Treatment
Number analyzed (Participants) | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 200
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 200
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 200
Nicotine Dependence - Cigarettes per day [Count of Participants; unit: Participants] — Nicotine Dependence was assessed at baseline using the The Fagerstrom Test for Nicotine Dependence (FTND); 6-item measure of nicotine dependence (cigarettes per day (CPD) and minutes to the first cigarette after waking).
  Participants
    <=10 | 74
    11-19 | 53
    >=20 | 70
    Refused to Answer | 3
Nicotine Dependence - Participants reported smoking their first cigarette with 5 minutes of walking [Count of Participants; unit: Participants] — Nicotine Dependence was assessed at baseline using the The Fagerstrom Test for Nicotine Dependence (FTND); 6-item measure of nicotine dependence (cigarettes per day (CPD) and minutes to the first cigarette after waking).
  Participants | 64
Demographics (Employment Status) [Count of Participants; unit: Participants] — Employment: self-reported employment status
  Participants
    Employed | 135
    Unemployed | 63
    Refused to Answer | 2
Demographics (Education) [Count of Participants; unit: Participants] — Education: self-reported years of education
  Participants
    < High School | 116
    High School/GED | 39
    Some College | 28
    Some kind of degree (Voc/AA/BS and up) | 16
    Refused to Answer | 1
Demographics (Household Income) [Count of Participants; unit: Participants] — Income: self-reported household income
  Participants
    <$12,000 | 30
    $12,001 - $30,000 | 68
    $30,001 - $54,000 | 54
    > $54,001/year | 20
    Refused to Answer | 28
Demographics (Spouse/Partner) [Count of Participants; unit: Participants] — Marital Status: self-report of participants with partner or no partner
  Participants
    No partner | 61
    Partner | 138
    Refused to Answer | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 24-Hour Smoking Abstinence (Week 3 Post Quit Day)
Description: Biochemically verified 24-hour point prevalence abstinence rates based on a completers-only approach.
Time Frame: Week 3 post quit day
Population: Completers-Only
Measure: Count of Participants; unit: Participants
Groups:
- Smoking Cessation Treatment: 6 wks of nicotine patch therapy, self-help guide and in-person/telephone individual counseling (6 sessions within 3 weeks of Quit date) based on Tobacco Use and Dependence Clinical Practice Guideline
Arm/Group | Smoking Cessation Treatment
Number analyzed (Participants) | 168
Participants | 100

2. Primary Outcome: 24-Hour Smoking Abstinence (Week 26 Post Quit Day)
Description: Biochemically verified 24-hour point prevalence abstinence rates based on a completers-only approach.
Time Frame: Week 26 post quit day
Population: Completers -only
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Treatment
Number analyzed (Participants) | 119
Participants | 41

3. Primary Outcome: 7-Day Smoking Abstinence (Week 3 Post Quit Day)
Description: Biochemically verified 7-day point prevalence abstinence rates based on a completers-only approach.
Time Frame: Week 3 post quit day
Population: Completers-only
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Treatment
Number analyzed (Participants) | 168
Participants | 76

4. Primary Outcome: 7-Day Smoking Abstinence (Week 26 Post Quit Day)
Description: Biochemically verified 7-day point prevalence abstinence rates based on a completers-only approach.
Time Frame: Week 26 post quit day
Population: Completers only
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Treatment
Number analyzed (Participants) | 119
Participants | 33

5. Primary Outcome: 30-Day Smoking Abstinence (Week 26 Post Quit Day)
Description: Biochemically verified 30-day point prevalence abstinence rates based on a completers-only approach.
Time Frame: Week 26 post quit day
Population: Completers only
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Treatment
Number analyzed (Participants) | 119
Participants | 28

6. Primary Outcome: 7-Day Smoking Abstinence (Week 3 Post Quit Day) Intent to Treat
Description: Biochemically verified 7-day point prevalence abstinence rates using an intent-to-treat approach
Time Frame: Week 3 post quit day
Population: Continuous Abstinence Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Treatment
Number analyzed (Participants) | 200
Participants | 57

7. Primary Outcome: 7-Day Smoking Abstinence (Week 26 Post Quit Day) Intent to Treat
Description: Biochemically verified 7-day point prevalence abstinence rates using an intent-to-treat approach
Time Frame: Week 26 post quit day
Population: Continuous Abstinence Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Treatment
Number analyzed (Participants) | 200
Participants | 20

8. Primary Outcome: 7-Day Smoking Abstinence (Week 3 Post Quit Day) Continuous Abstinence
Description: Biochemically verified 7-day point prevalence abstinence rates using a completers-only approach
Time Frame: Week 3 post quit day
Population: Continuous Abstinence Completers-only
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Treatment
Number analyzed (Participants) | 168
Participants | 57

9. Primary Outcome: 7-Day Smoking Abstinence (Week 26 Post Quit Day) Continuous Abstinence
Description: Biochemically verified 7-day point prevalence abstinence rates using a completers-only approach
Time Frame: Week 26 post quit day
Population: Continuous Abstinence Completers-only
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Treatment
Number analyzed (Participants) | 119
Participants | 20

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline up to 26 weeks
Arm/Group | Smoking Cessation Treatment
All-Cause Mortality (participants affected / at risk) | 0/200
Serious Adverse Events (participants affected / at risk) | 0/200
Other Adverse Events (participants affected / at risk) | 0/200

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes